CLINICAL TRIAL: NCT02596100
Title: A Bioequivalence Study to Compare the Pharmacokinetics of Two Betrixaban Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Portola Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 15-020
Record Dates: First submitted 2015-10-21; First posted 2015-11-04 (Estimated); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Healthy
Keywords: Bioequivalence
MeSH Terms: interventions — betrixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tablet (Experimental): 80mg immediate release tablet
  Interventions: Drug: Betrixaban
- Capsule (Experimental): 80mg immediate release capsule
  Interventions: Drug: Betrixaban

INTERVENTIONS:
Drug: Betrixaban

SUMMARY:
This is a single center open label randomized 4-period 2-sequence replicated crossover design study. A total of 52 healthy subjects will be randomized.

DETAILED DESCRIPTION:
Serial blood samples will be obtained for PK evaluation.

ELIGIBILITY:
Inclusion Criteria:

* All inclusion criteria must be satisfied within 30 days of enrollment and must be documented in the source documents.
* A healthy man or woman between the ages of 18 and 60
* Has no clinically significant findings in medical history, physical examination, EKG and vital signs
* Weighs > 45 kg (99 lbs.) and has body mass index (BMI) < 30 kg/m2
* Agrees to abstain from alcohol consumption for 48 hrs prior to dosing and for the duration of each of the study in-house periods
* Is a non-smoker or light smoker (no more than the equivalent of five cigarettes per day) and agrees to abstain from smoking for the duration of each of the study in-house periods

Exclusion Criteria:

* None of the exclusion criteria may be present for enrollment
* Known history (including family history) or symptoms of any clinically significant bleeding (i.e. a bleeding that required medical attention) or a vascular malformation
* Major surgery, severe trauma or bone fracture within 3 months of the first dose of the study drug or a planned surgery within 1 month after the last dose of the study drug
* History of blood donation of more than 500 mL within 3 months prior to the first dose of the study drug
* History of alcohol abuse (greater than 3 alcoholic beverages per day)
* Positive screen for drugs of abuse
* Positive serology test for HIV, Hepatitis B or C
* Has any allergy or sensitivity to fXa inhibitors

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence analysis using total area under the curve (Total AUC) after a single dose of Betrixaban in healthy subjects | 120 hours
Bioequivalance analysis using peak concentration in plasma (Cmax) after a single dose of Betrixaban in healthy volunteers | 120 hours